CLINICAL TRIAL: NCT00111774
Title: An Open Label Phase 2 Clinical Trial to Evaluate the Safety and Efficacy of ABX-EGF in Patients With Metastatic Colorectal Carcinoma
Brief Title: Evaluating ABX-EGF in Patients With Metastatic ColorectalCarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20025405
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer; Carcinoma
Keywords: Colon Cancer, Rectal Cancer; Colorectal Carcinoma, EGFr; Metastatic Cancer, ABX-EGF; Panitumumab, Abgenix; Clinical Trial, Immunex, Amgen; Metastatic Colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis | interventions — Panitumumab

INTERVENTIONS:
Drug: ABX-EGF

SUMMARY:
The purpose of this study is to determine if ABX-EGF is safe and efficacious in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria: Cohort A: - Pathologic diagnosis of colorectal carcinoma fine needle aspiration or tissue biopsy - Metastatic colorectal carcinoma - Must have previously failed therapy with a fluoropyrimidine and either irinotecan or oxaliplatin; may have received both irinotecan and oxaliplatin; chemotherapeutic agents may have been given concurrently or sequentially. - May have received prior radiotherapy (target lesions should not have been irradiated) - Bidimensionally measurable disease - Paraffin-embedded tumor tissue available for immunohistochemistry (IHC) studies of epidermal growth factor receptor (EGFr) expression (archived tissue is acceptable) - Tumor-expressing EGFr by immunohistochemistry (staining must be 2+ or 3+ in greater than or equal to 10% of evaluated tumor cells; staining and evaluation to be conducted at a central laboratory) - ECOG score of 0 or 1 - Adequate hematologic, renal, and hepatic function Cohort B: - The same inclusion criteria from Cohort A will apply to Cohort B, with the exception of the following tumor expressing EGFr criterion:

*Cohort B will include subjects who have IHC staining of 1+ present in greater than 10% evaluated tumor cells, OR IHC staining of the sum of 1+, 2+ and 3+ present in greater than 10% evaluated tumor cells but with the sum of 2+ and 3+ present in less than 10% evaluated tumor cells Exclusion Criteria: Cohorts A and B: - Female subject (e.g., of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized or not abstinent) who is not willing to use an oral or implanted contraceptive, double barrier birth control, or an intrauterine device (IUD) during the course of the study and for 6 months following the last ABX-EGF infusion - Female subject who is breast feeding or who has a positive serum pregnancy test within 72 hours prior to the first ABX-EGF infusion - Male subject who is not willing to use adequate contraception upon enrollment into this study and for 1 month following the last ABX-EGF infusion - Untreated brain metastases - Use of systemic chemotherapy or radiotherapy within 30 days prior to the first dose of ABX-EGF - Chemotherapy other than fluoropyrimidines, irinotecan or oxaliplatin for colorectal carcinoma. Leucovorin and levamisole are not considered as chemotherapy in this exclusion criterion. - Prior EGFr targeting agents - Prior investigational drugs with potential antitumor activity (experimental small molecules within 30 days prior to the first ABX-EGF infusion, experimental proteins/antibodies within 3 months prior to the first ABX-EGF infusion) - If prior history of cancer, other than colorectal carcinoma, basal cell carcinoma, or cervical carcinoma in situ, no treatment or active disease within 5 years - Myocardial infarction within past year - Left ventricular ejection fraction (LVEF) less than 45%, as measured by multiple-gated acquisition (MUGA) scan - Known to be HIV positive - History of any chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation or study drug administration or may interfere with the interpretation of study results - Subject allergic to the ingredients of the study medication or to Staphylococcus Protein A - Unwilling or unable to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-03

PRIMARY OUTCOMES:
To assess Objective Response at Week 8 of Cycle 1

SECONDARY OUTCOMES:
To evaluate additional measures of the clinical efficacy of ABX-EGF in subjects with metastatic colorectal carcinoma. (progression free survival, survival time, best overall response, and time to disease progression)
To determine the safety of ABX-EGF in subjects with metastatic colorectal carcinoma. (incidence of AEs, laboratory abnormalities, and other safety parameters)
To evaluate the safety and efficacy of ABX-EGF in subjects with lower tumor epidermal growth factor receptor (EGFr) expression

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Hecht JR, Patnaik A, Berlin J, Venook A, Malik I, Tchekmedyian S, Navale L, Amado RG, Meropol NJ. Panitumumab monotherapy in patients with previously treated metastatic colorectal cancer. Cancer. 2007 Sep 1;110(5):980-8. doi: 10.1002/cncr.22915. PMID 17671985
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com